CLINICAL TRIAL: NCT01176045
Title: Measurement of Refractive Surgery Induced Dry Eye Using Tear Osmolarity Testing
Brief Title: TearLab Refractive Surgery Dry Eye Study
Status: Completed | Type: Observational
Sponsor: TearLab Corporation (Industry)
Collaborators: TLC Laser Eye Center (Unknown); Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Other Study IDs: TP00087
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye Disease; Osmolarity; Refractive Surgery; Lasik; TearLab
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-surgical treatment: Patients who are pre & post-surgical treated with ocular lubricants.
- Non-presurgical treatment: Patients who are only post-surgical treated with ocular lubricants

SUMMARY:
The primary objective of this study is to determine how pre & post-operative tear osmolarity levels relate to rates of dry eye symptoms related to refractive surgery and if differences exist in patients who are pre-treated with ocular lubricants vs. those treated only post-operatively.

DETAILED DESCRIPTION:
Dry eye disease is a common and major source of disability, whether occurring as a primary disorder or as a component of other diseases and its onset may be triggered or modified by exposure to systemic drugs, contact lens wear, ocular surgery and adverse environmental and work conditions. The development of a reliable, highly sensitive and specific test for the clinical diagnosis of dry eye is a major unmet clinical need, particularly to differentiate it from common conditions such as ocular allergy which exhibit similar presenting symptoms. Tear hyper-osmolarity is central to the dry eye disease process and the measurement of tear osmolarity could serve not only as a highly accurate diagnostic test but also as a measure of disease severity and a means to monitor treatment efficacy.

Recently, there have been reports in the literature regarding dry eye disease; both early and chronic following refractive surgery, with many cases potentially being previously inadvertently undiagnosed dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, twenty-one years of age or older.
* Confirmed diagnosis of refractive error receiving LASIK surgery.
* Patient motivation and willingness to cooperate with the investigator and ability to return for all visits during the study.

Exclusion Criteria:

* Compromised cognitive ability that may be expected to interfere with study compliance.
* Clinically significant eyelid deformity or eyelid movement disorder that is caused by conditions such as notch deformity, incomplete lid closure, entropion, ectropion, hordeola or chalazia.
* Previous ocular disease leaving sequelae or requiring current topical eye therapy other than for DED, including, but not limited to: active corneal or conjunctival infection of the eye and ocular surface scarring.
* Active ocular allergy
* Patients requiring punctual occlusion prior to surgery
* Patients requiring cyclosporine ophthalmic emulsion prior to surgery
* Standard exclusion criteria for refractive surgery used by each surgeon.
* Known hypersensitivity to any of the agents used in testing
* Ophthalmologic drop use within 2 hours of any visit

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo refractive surgery with no previous diagnosis of dry eye disease.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Relation of pre & post-operative tear osmolarity levels to dry eye and dry eye symptoms in refractive surgery | 6 months post surgery

SECONDARY OUTCOMES:
To determine if differences exist in patients who are pre-treated with ocular lubricants vs. those treated only post-operatively | 6 months post-surgical
To determine if tear osmolarity levels relate to visual acuity outcomes related to refractive surgery | 6 months post-surgical

CONTACTS AND LOCATIONS:
Overall Officials: James Owen, OD, Study Director — TLC The Laser Eye Center
Locations (8):
- United States (8):
  - Connecticut TLC, Fairfield, Connecticut
  - Westchester TLC, Westchester, Illinois
  - Oklahoma City TLC, Oklahoma City, Oklahoma
  - Tulsa TLC, Tulsa, Oklahoma
  - Kremer Eye Center, King of Prussia, Pennsylvania
  - San Antonio TLC, San Antonio, Texas
  - Salt Lake City TLC, Salt Lake City, Utah
  - Reston TLC, Reston, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Study data has been shared in Vienna 2011. Patients with pre-operative hyperosmolarity (≥ 308 mOsms/L) demonstrated worse long-term uncorrected visual acuity. An abnormal tear film may cause inaccurate wavefront aberrometry. For patients with preoperative osmolarity ≥ 308 mOsms/L, it may be important to continue therapy for at least 3 months. Similarly, surgeons should measure tear osmolarity preoperatively as staining was too insensitive to identify at-risk patients. Patients treated pre-operatively with AMO Blink® Tears achieved normal osmolarity faster than those untreated before surgery.